CLINICAL TRIAL: NCT02813902
Title: A Pilot Trial of Polypodium Leucotomos in Preventing Skin Cancer and Its Precursors
Brief Title: A Trial of Polypodium Leucotomos in Preventing Skin Cancer and Its Precursors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of funding.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Maryam M Asgari, Director, Dermatology High Risk Skin Cancer Clinic, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2016P001176
Record Dates: First submitted 2016-06-07; First posted 2016-06-27 (Estimated); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Keratosis, Actinic; Keratosis; Skin Neoplasms
MeSH Terms: conditions — Keratosis, Actinic; Keratosis; Skin Neoplasms | interventions — Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heliocare (Active Comparator): 240 mg administered orally daily
  Interventions: Drug: Heliocare with Fernblock PLE technology
- Sugar pill (Placebo Comparator): a sugar pill matching the Heliocare tablet in look and weight will be administered orally daily
  Interventions: Other: Sugar Pill

INTERVENTIONS:
Drug: Heliocare with Fernblock PLE technology — 240 mg taken orally daily over the course of 1 year
  Other Names: Polypodium leucotomos extract capsules
  Arms: Heliocare
Other: Sugar Pill — A pill that appears similar to the supplement
  Other Names: Placebo
  Arms: Sugar pill

SUMMARY:
This proposal describes a pilot study to gather preliminary evidence of efficacy, tolerability and toxicity of oral PLE among a high-risk skin cancer population for the prevention of Actinic keratosis (AKs) and keratinocytes (KCs) to gain insight into optimal methods for recruitment, intervention development, data collection, and promoting protocol adherence prior to conducting a fully powered trial. The primary clinical outcome is AKs as measured by a clinical dermatologist, with skin cancer as a secondary clinical outcome. The investigators will also assess histologic markers of Ultra Violet (UV) damage, which have previously been shown to be reduced with oral PLE use in human studies, namely formation of UV-induced cyclo pyrimidine dimer positive cells and number of sunburn cells among epidermal keratinocytes. Results generated from this proposal will form the foundation of a fully powered clinical trial of the effect of PLE on the risk of AKs and KCs. The results may also provide information about this promising dietary supplement which may provide extra protection for a high-risk skin cancer population.

DETAILED DESCRIPTION:
Polypodium leucotomos is a tropical fern, the extract of which has shown photoprotective effects in animal and human models, and is currently available as an over-the-counter dietary supplement. Polypodium leucotomos extract (PLE) has been shown in laboratory, animal, and clinical studies to serve as a potent antioxidant that helps mitigate UV-induced damage by scavenging free radicals and reactive oxygen species. Oral consumption of PLE in human studies has been shown to significantly reduce the number if UV-induced sunburn cells and DNA damage, and to inhibit photosensitization. Importantly, PLE appears to be exceptionally well-tolerated with no serious reported adverse side effects.

PLE has been studied in numerous trials for many conditions, including skin diseases. Doses up to 1200 mg per day have been used in clinical studies, though doses for prevention of sun-damage are typically in the range of 480 mg per day. To date, no serious adverse effects have been clearly attributed to the use of PLE (this high tolerability is one of the reasons for the great interest in the clinical use of PLE). Oral consumption of other fern species, such as Polypodium vulgare, have been associated with low blood pressure and increased heart rate. On theoretical grounds, similar side effects may be possible with PLE.

ELIGIBILITY:
Inclusion Criteria:

* Must be male or female and at least 18 years of age.
* Female patients must be of:

  * Non-childbearing potential;
  * Childbearing potential, provided negative urine pregnancy test and using effective contraception.
* Dermatologist-rendered diagnosis of AK in the past 2 years.

Exclusion Criteria:

* History of >2 skin cancers in the past 5 years
* History of dementia
* Cardiovascular disease, defined as Blood Pressure (BP) <90/60 or Heart rate (HR) >110 in the past year or a history of myocardial infection
* Inflammatory bowel disease/irritable bowel syndrome
* Treatment with Fluorouracil, imiquimod, diclofenac, or photodynamic therapy in the past 8 weeks
* Intention to seek more aggressive AK therapy such as photodynamic therapy, laser surgery in next 12 months
* Serious psychological illness
* History of alcohol or drug abuse
* Any disease or condition which would interfere with study participation or unduly increase risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Total number of new clinically visable AKs as measured by a full skin exam performed by a blinded, board certified dermatologist (Dr. Asgari). | one year

SECONDARY OUTCOMES:
Histologic presence of UV-induced cyclobutane pyrimidine dimer positive cells | one year
Degree of solar elastosis assessed using Verhoeff stain on biopsy specimens obtained from punch biopsy | one year
Counts of sunburnt cells in sun exposed skin | one year

CONTACTS AND LOCATIONS:
Overall Officials: Maryam M Asgari, MD, MPH, Principal Investigator — Massachusetts General Hospital